CLINICAL TRIAL: NCT01182610
Title: A Phase II Study of Pre-operative Panitumumab, Paclitaxel, Carboplatin and Continuous Infusion 5FU in the Treatment of Potentially Resectable Gastroesophageal Adenocarcinoma
Brief Title: Panitumumab, Paclitaxel, Carboplatin and 5FU in the Treatment of Potentially Resectable Gastroesophageal Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety concern in a similar trial enrolling the same patient population
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACORN ARCHESO0611
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Results first posted 2012-11-28 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Gastroesophageal Adenocarcinoma; Adenocarcinoma of the Distal Esophagus; Adenocarcinomas of the Gastroesophageal Junction; Adenocarcinoma of the Proximal Stomach
MeSH Terms: interventions — Panitumumab; Paclitaxel; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Panitumumab 9mg/kg on Days 1, 22, and 43
  Paclitaxel 200mg/m2 on Days 1 and 22
  Carboplatin AUC=6 on Days 1 and 22
  5FU 225mg/m2/day on Days 1-15 and 22-36
  Interventions: Drug: Panitumumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: 5FU

INTERVENTIONS:
Drug: Panitumumab — Panitumumab 9mg/kg on Days 1, 22, and 43
  Other Names: Vectibix
Drug: Paclitaxel — Paclitaxel 200mg/m2 on Days 1 and 22
  Other Names: Taxol
Drug: Carboplatin — Carboplatin AUC=6 on Days 1 and 22
  Other Names: Paraplatin, CBDCA
Drug: 5FU — 5FU 225mg/m2/day on Days 1-15 and 22-36
  Other Names: 5-fluorouracil

SUMMARY:
This is an open-label, Phase II, single-stage study evaluating the use of panitumumab, paclitaxel, carboplatin and 5FU as an induction regimen in subjects with gastroesophageal adenocarcinoma. The expectation is that this combination will both increase potential overall survival by incorporating novel biologic therapy in the neoadjuvant setting and decrease potential surgical mortality by eliminating pre-operative radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven adenocarcinoma of the distal esophagus, gastroesophageal junction, or proximal stomach (within 5cm of gastroesophageal junction)
* No prior treatment for this disease
* AJCC (American Joint Committee on Cancer) clinical stage II to IVA, potentially resectable disease
* Measurable disease per RECIST 1.0 criteria
* Medically fit for surgery; surgical consultation is encouraged prior to initiation of treatment
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1
* Male or female; aged equal to or greater than 18 years
* Life expectancy of greater than 3 months
* Good organ, metabolic, bone marrow, and pulmonary function as specified in the protocol
* Functioning central venous access device prior to treatment initiation
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for at least 6 months following the last administration of panitumumab
* Ability to understand and the willingness to sign a written IRB (Institutional Review Board) approved informed consent

Exclusion Criteria:

* Prior treatment for this disease
* History of another primary cancer except curatively treated in situ cervical cancer, curatively resected nonmelanoma skin cancer, or other primary solid tumor curatively treated with no active disease present and no treatment administered for at least 5 years prior to enrollment
* History or known presence of central nervous system metastases
* History of allergic reactions attributed to compounds similar chemical or biologic composition to panitumumab, paclitaxel, carboplatin, or 5FU
* Prior anti-EGFr-antibody therapy or treatment with small molecule EGFr inhibitors
* Systemic chemotherapy, hormonal therapy, immunotherapy, or experimental or approved proteins/antibodies within 30 days prior to enrollment
* Chronic use of immunosuppressive agents with the exception of corticosteroids
* Any investigational agent or therapy within 30 days prior to enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of interstitial lung disease, e.g., pneumonitis or pulmonary fibrosis or any evidence of interstitial lung disease on baseline chest CT scan
* History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with study participation or investigational product(s) administration or may interfere with the interpretation of the results
* Unwilling or unable to comply with study requirements
* Female who tests positive for serum or urine pregnancy test or is breast feeding
* Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, acute or chronic active hepatitis B infection
* Major surgery within 28 days or minor surgery within 7 days prior to treatment. Placement of a central venous access device less than one day prior to treatment start
* Male or female of childbearing potential (women who are post-menopausal less than 52 weeks, not surgically sterilized, or not abstinent) not consenting to use adequate contraception prior to study entry and for at least 6 months following the last administration of panitumumab
* Arterial ischemic event (myocardial infarction, stroke) within 3 months prior to enrollment
* Ongoing therapeutic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hermann, MD, Principal Investigator — Accelerated Community Oncology Research Network
Locations (1):
- Clopton Clinic, Jonesboro, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 sites associated with Accelerated Coummunity Oncology Research Network, Inc. (ACORN) or Georgia Center for Oncology Research and Education (GA-CORE)participated in this study. Enrollment started in May 2011 and was closed in November 2011 due to toxicities observed in a similar trial.
Pre-assignment Details: Informed consent was obtained from the subject. The Subject underwent a screening period of up to 35 days during which pre-study assessments were completed.
Groups:
- Treatment Group: Treatment group : Panitumumab 9mg/kg on Days 1, 22, and 43
  Paclitaxel 200mg/m2 on Days 1 and 22
  Carboplatin AUC=6 on Days 1 and 22
  5FU 225mg/m2/day on Days 1-15 and 22-36
Period: Overall Study
Arm/Group | Treatment Group
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Panitumumab 9mg/kg on Days 1, 22, and 43
  Paclitaxel 200mg/m2 on Days 1 and 22
  Carboplatin AUC=6 on Days 1 and 22
  5FU 225mg/m2/day on Days 1-15 and 22-36
  Treatment group : Panitumumab 9mg/kg on Days 1, 22, and 43
  Paclitaxel 200mg/m2 on Days 1 and 22
  Carboplatin AUC=6 on Days 1 and 22
  5FU 225mg/m2/day on Days 1-15 and 22-36
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 73 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The primary endpoint is overall response rate (ORR) as determined per RECIST guidelines version 1.1 from baseline and restaging scans conducted between Days 36 to 43. Response is defined as the occurrence of either Complete Response (CR) or Partial Response (PR) as best response. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. A PR is defined as at least a 30% decrease in the sum of diameters of the target lesions taking as reference the baseline sum diameters.
Time Frame: From the start of study treatment until restaging evaluation performed between days 36 to 43
Population: This study was closed due to a notification letter (November 1, 2011) and preliminary results from another trial that included panitumumab as part of combination chemotherapy for gastroesophageal cancer. The study was closed by mutual consent from the Principal Investigator, Sponsor, and Funder.
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

2. Secondary Outcome: Pathologic Response Rate
Description: The patient will be scored as having had a pathologic complete response (pCR) if the routine histologic examination of the resected specimen shows no residual invasive cancer by standard hematoxylin and eosin (H&E) examination.
Time Frame: At time of surgery (between days 50 to 64)
Population: as for outcome 1
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Resection Rate of Surgery
Description: The patient will be scored as having an R0 resection, if no invasive cancer is detected involving the margins of the resection by routine microscopic hematoxylin and eosin (H&E)examination, and the operative report indicates complete resection with no residual disease.
  The patient will be scored as having an R1 resection, if invasive cancer is detected involving the margins of resection by routine microscopic hematoxylin and eosin (H&E) examination, and the operative report indicates complete resection with no residual disease.
  The patient will be scored as having an R2 resection, if the operative report indicates incomplete resection or gross residual disease.
Time Frame: At time of surgery (between days 50 to 64)
Population: as for outcome 1
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Thirty-day Surgical Mortality
Description: All subjects who have undergone surgical resection will be followed for a 30-day postoperative safety evaluation. Death from any cause within 30 days of the date of surgery will be considered a surgical mortality death.
Time Frame: From date of surgery to 30 days after date of surgery
Population: as for outcome 1
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

5. Secondary Outcome: Survival
Time Frame: 2-year survival from first dose of panitumumab
Population: as for outcome 1
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected beginning on day 1 of study treatment through the End of Treatment visit (30 days post-operative, 6 weeks from last treatment administration if treatment failure, or 30 days from last dose of study treatment if early withdrawal).
Description: Systematic Assessment- subjects were assessed for adverse events on day 1 of each cycle by either the research coordinator, treating physician, or other appropriate sub-investigator.
Groups:
- Treatment Group: Panitumumab, Paclitaxel, Carboplatin and 5FU: Panitumumab 9mg/kg on Days 1, 22, and 43; Paclitaxel 200mg/m2 on Days 1 and 22; Carboplatin AUC=6 on Days 1 and 22; 5FU 225mg/m2/day on Days 1-15 and 22-36
Arm/Group | Treatment Group: Panitumumab, Paclitaxel, Carboplatin and 5FU
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group: Panitumumab, Paclitaxel, Carboplatin and 5FU (N=1)
Neutropenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Mucosal inflammation (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group: Panitumumab, Paclitaxel, Carboplatin and 5FU (N=1)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abnormal sensation in eye (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Generalised oedema (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Pyrexia (General disorders) | 1
Weight Decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Depressed level of consiciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This study was closed due to notification and preliminary results from a trial including panitumumab as part of combination chemotherapy for gastroesophageal cancer. The study was closed by mutual consent from the PI, Sponsor, and Funder.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication or presentation of Sponsored Research results, Researcher agrees to provide Amgen 60 days to review a manuscript and 15 days to review any poster presentation, abstract or other written or oral materials derived from a Study. If Amgen requests in writing, the Researcher shall withhold material an additional 60 days. Amgen reserves the right to remove confidential information from any publications. The Researcher shall reference Amgen's support of the Study in any material.